CLINICAL TRIAL: NCT03967418
Title: Study BANCO2: Behavioral Addictions and Related NeuroCOgnitive Aspects : Monocentric, Prospective, Controlled, Open-label Study Conducted With a Sample of Patients With Behavioural Addiction
Brief Title: Behavioral Addictions and Related NeuroCOgnitive Aspects
Acronym: BANCO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC19_0177
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Behavioral Addiction
Keywords: Behavioral addiction; neurocognition; neuropsychology; sexual addiction; eating disorders
MeSH Terms: conditions — Compulsive Sexual Behavior Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with behavioral addictions (Other): Patients suffering from behavioural addiction (sexual addiction and eating disorders with bulimia episodes) will be recruited
  Interventions: Behavioral: Cognitive and clinical assessment
- Healthy volunteers (Other): Healthy volunteers will be matched on gender, age and education level to patients
  Interventions: Behavioral: Cognitive and clinical assessment

INTERVENTIONS:
Behavioral: Cognitive and clinical assessment — The content of the assessment will be the same for all subjects and will consist of a cognitive assessment (neurocognition, social cognition, metacognition, emotional reactivity) and a clinical assessment (impulsivity, personality, psychiatric and addictive comorbidities)

SUMMARY:
Improving knowledge about behavioural addictions is a real public health issue. The etiopathogenic model of behavioural addictions is multifactorial, with various risk and vulnerability factors, involved in the initiation and maintenance of the disorders. Among these factors, neurocognitive alterations associated with behavioural addictions has recently aroused interest among researchers.

To our knowledge, there is no work wich compared several behavioural addictions with each other on a neurocognitive level. Moreover, neurocognitive data concerning certain behavioural addictions (such as sexual addiction) is almost non-existent. However, understanding the neurocognitive profiles of these patients would allow the investigators, on the one hand, to reinforce the existing literature and improve our understanding of the global process of addiction, and on the other hand, to propose alternative approaches to its management, taking into account the neurocognitive difficulties of the patients.

The investigators therefore propose to explore the neurocognitive alterations of patients suffering from several behavioural addiction (sexual addiction and eating disorders with bulimia episodes), by comparing them with each other, to matched healthy control groups and to a recognized behavioural addiction (gambling disorder; data from the BANCO study - NCT03202290).

ELIGIBILITY:
Inclusion Criteria for all participants:

* More than 15 years and 3 months old
* Mastering the French language
* Social Security Affiliates
* Having given consent
* Correct level of vision allowing the reading of instructions, the distinction of shapes and colours and the understanding of shapes and images presented in cognitive tasks (subjectively attested by the patient)
* Correct hearing level, allowing a good understanding of the sounds presented (subjectively attested by the patient and the assessor at the first contact for eligibility)

Inclusion criteria for patients:

* Suffering from one of the behavioural addiction explored
* Beginning treatment in the Addictology department of the University Hospital of Nantes

Inclusion criteria for healthy volunteers:

- Free from the explored behavioural addictions

Exclusion Criteria for all participants:

* Current and not stabilized psychiatric and addictive disorders (mood disorders, anxiety disorders and substance-use disorders except nicotine, lifetime psychotic syndrome), diagnosed by the MINI and after consultation with the clinician,
* Non stabilized endocrine disorders
* Neurological disorders (such as head trauma, neurodegenerative diseases, unbalanced epilepsy, mental retardation, etc.),
* Taking a psychotropic treatment wich is not stabilized for at least 2 weeks,
* Consumption of a psychoactive substance - other than nicotine - within the 12 hours prior to the assessment,
* Color blindness
* Cardiac problems self-reported by the patient, in order to avoid bias in the measurement of cardiac parameters,
* Electrical implants as declared by the participant (to avoid measurement artifacts)
* Having benefited from current or past cognitive remediation program
* Reporting being pregnant or breastfeeding
* Current participation or in the past month in a pharmacological research protocol
* Presenting difficulties for reading or writing French
* Being under guardianship
* With significant cognitive impairment not compatible with de cognitive assessment

Exclusion criteria for healthy volunteers :

- Suffering from one of the behavioural addiction explored

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Scores obtained at the various neurocognitive tests used | 4 hours
  A composite score will be created to reflect the overall level of cognitive performance of individuals with behavioral addictions, compared to healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Marie GRALL BRONNEC, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hurel E, Grall-Bronnec M, Thiabaud E, Saillard A, Hardouin JB, Challet-Bouju G. A Case-Control Study on Behavioral Addictions and Neurocognition: Description of the BANCO and BANCO2 Protocols. Neuropsychiatr Dis Treat. 2021 Jul 20;17:2369-2386. doi: 10.2147/NDT.S292490. eCollection 2021. PMID 34321880